CLINICAL TRIAL: NCT04141956
Title: Incidence of Use of High-Flow Nasal Cannula Oxygen Therapy in Intensive Care Units : Prospective, Multi-center, Epidemiological, Uncontrolled Study
Brief Title: Incidence of Use of High-Flow Nasal Cannula Oxygen Therapy in Intensive Care Units Patients
Acronym: OHE-REA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0386
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High-Flow Nasal Cannula — Incidence of nasal High Flow Nasal Cannula (HFNC) Oxygen therapy in patients admitted to intensive care.

SUMMARY:
Patients with one or more organ failure (heart, lung) require hospitalization in intensive care where these failures can be managed. Nearly 30% of patients in intensive care units are hospitalized for acute respiratory distress (lung failure). This failure occurs in about 20% of postoperative patient, but it can also occur in the context of a pathology specific to the lung or after weaning of mechanical ventilation.

It is therefore interesting to develop several techniques to provide oxygen to these patients with the aim in particular to avoid the use of intubation (insertion of a tube into the trachea to achieve artificial ventilation). For the past ten years, High-Flow Nasal Canula (HFNC) has developed. This technique reduces the need for intubation but the studies are contradictory, however they agree on its ease of use and the few risks associated with it. The principle of this technique is to deliver a humidified and heated gas mixture at a high rate through large nasal cannula. The advantage of this device is its non-invasive and the possibility of administering a large amount of oxygen. There is a certain craze for this oxygenation technique despite few scientific studies in the literature. However, it requires the expertise of the medical and paramedical team so as not to delay intubation.

The investigators propose to carry out an observational study (without any modification of the usual practices) with epidemiological aim in order to make an inventory of the modes of use of the HFNC, in particular on its frequency of use and on its duration of use per patient hospitalized in intensive care. The investigators will recruit all HFNC patients in intensive care units (20 centers) (30 patients / center): 15 after weaning of mechanical ventilation and 15 others for other reasons. Patients will be followed every day and up to 48 hours after removal of the HFNC.

DETAILED DESCRIPTION:
Oxygen therapy is one of the most prescribed treatments in medicine, especially in intensive care patients. It is an adjuvant therapy as a respiratory support whose goal is to maintain optimal ventilation and oxygenation and to improve alveolar gas exchange. HFNC is in full swing and increasingly used as an alternative to standard oxygen therapy in patients with acute respiratory failure (ARF). This nasal oxygenation technique, humidified and heated at high flow, initially developed in pediatrics is a simple and effective alternative for adults in IRA hospitalized in intensive care. The OHD makes it possible to deliver a gas mixture with a maximum flow rate of 70 l/min of oxygen via a generator connected to a chamber for humidifying and heating gases at 37 °. OHD offers several physiological benefits that could encourage its use: administration of a high oxygen-inspired fraction (FiO2), generation of a low level of flow-dependent PEP, reduction of nasopharyngeal resistance, and wash-rinse of the anatomic dead space, thanks to the high nasal flow. It is also a comfortable technique compared to the NIV.

This means of oxygen therapy is increasingly used in routine practice in our patients admitted to intensive care for non-hypercapnic respiratory insufficiency, especially since this reason for admission represents approximately 30% of our patients. HFNC is interesting because of the pathophysiological advantages mentioned above, especially in patients with ARI who are hypoxemic. These patients have a greater respiratory work with an increase in inspiratory flow of up to 30-40l/min on average and exceed 60l/min or 120l/min. This flow rate can not be compensated by conventional oxygen therapy, limited to 15 l / min, which is insufficient to guarantee a constant and high oxygen concentration during inspiration, hence the interest of OHD capable of delivering a maximum flow rate of 70 l/min.

Its use has grown exponentially since 2015, the year of publication of the multicenter study FLORALI, comparing different methods of oxygen therapy (OHD vs conventional oxygen therapy vs NIV / OHD) in 310 patients with acute non-hypercapnic respiratory failure (2). In this study, the primary endpoint is the rate of intubation. There was no significant difference (p = 0.17) between the 3 techniques used: OHD (37.7%), conventional oxygenation (46.8%) and VNI / OHD (50%), despite a clear decrease in mortality at J90 (p = 0.02) in the OHD group (12%) compared to the other 2 strategies but this is a secondary endpoint. However, in the most hypoxemic patients (P / F ≤ 200), post-hoc analysis found a significantly lower intubation rate (p = 0.009) in patients treated with OHD alone (35%) compared with conventional oxygen therapy group (53%) and NIV / OHD (58%), with the same observation regarding the number of days without mechanical ventilation. These authors also published a post-hoc analysis of this study. They analyzed the effect of OHD in 82 immunocompromised patients and concluded that OHD patients had a better prognosis compared to those treated with conventional oxygen therapy or NIV. They found a significantly lower intubation rate (p = 0.04) in the HFNC group (31%) compared to conventional oxygen therapy (43%) and NIV (65%). These results should be interpreted with caution since Lemiale et al., In a large multicenter randomized study, did not show a significant difference in morbidity-mortality intubation in 374 immunosuppressed IRA patients treated with NIV (HFNC alone or NIV / HFNC) or standard oxygen therapy. These results are interesting, although they are post-hoc analyzes and secondary judgment criteria. A multicenter French randomized study was published recently and confirms the results of the Lemiale team (HFNC is no better than standard oxygen therapy in immunocompromised patients). For these patients, another multicenter randomized controlled French trial is underway (NCT02978300).

Currently more and more patients, admitted for non-hypercapnic ARF, are treated with HFNC in first intention as well as post-extubation, because of its pathophysiological advantages, its comfort and its simplicity of setting up and use, despite the result of a single multicenter randomized study, positive only on secondary endpoints and post-hoc analyzes.

In addition, a recent meta-analysis, by Corley et al., Of randomized studies on the use of HFNC concluded in an insufficient level of evidence to recommend HFNC in ARF patients with a risk of delayed intubation of these patient. It should be noted, however, that the studies analyzed are heterogeneous in terms of patients, mode of administration of HFNC and etiology of ARF. Some authors are interested in parameters such as the ROX index to target patients at risk or not to progress to intubation in patients treated with HFNC which would secure its use and guide clinicians. Studies are underway to investigate the benefit of this device in patients with chronic respiratory failure admitted for hypercapnic ARF compared to standard oxygen between NIV sessions (NCT03406572). These authors also published a study concerning the use of HFNC in pre-oxygenation compared with BAVU and demonstrated a decrease in desaturation in pre-intubation. However, other authors have moderated these results in another randomized study with a different methodology, especially in terms of the use of OHD in apneic oxygenation (absence of mandibular sub-luxation). These results still show the heterogeneity of the practices as for its use in pre intubation.

Regarding its use in weaning mechanical ventilation, HFNC is increasingly used especially in post-operative without real benefit proven in the literature.

For example, in the University Hospital of Nantes in the Intensive Resuscitation Medicine (ICU) department, in 2017, 110 patients in ARF, were treated by HFNC out of 191 patients admitted for IRA, or 58% (institutional figures). There is a certain craze for this oxygenation technique in intensive care despite the low level of evidence, hence the interest of our epidemiological study.

It is a prospective, observational, multicentric (20 centers), epidemiological French study whose main objective is to evaluate the incidence of HFNC use. In order to calculate the incidence of use of the HFNC, The investigators will ask the different centers to provide us with the number of patients hospitalized in intensive care during the period of inclusion. the secondary objectives are: evaluation of morbidity and mortality in intensive care: intubation rate, weaning failure, weaning mode of HFNC. Epidemiological data: modalities of use, duration of use and indications.

ELIGIBILITY:
Inclusion Criteria:

* all adults' patients, admitted to intensive care units treated with HFNC (indication is to discretion of doctor).

Exclusion Criteria:

* HFNC use for Preoxygenation and Apneic Oxygenation for Intubation
* Minor patient, adult patient under guardianship, protected persons, pregnant woman, prior inclusion in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults' patients, admitted to intensive care units treated with HFNC (indication is to discretion of doctor).
  For example : Acute Hypoxemic Respiratory Failure, Postoperative Respiratory Failure or systematic when weaning mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of nasal High-Flow Nasal Cannula (HFNC) Oxygen therapy in patients admitted to intensive care | 28 days after enrollment
  Incidence defined by: the ratio of the number of patients under HFNC on the number of patients admitted to intensive care during the period of inclusion.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Chu Jean Minjoz Besancon, Besançon
  - CHU CAEN, Caen
  - Polyclinique Du Cotentin, Cherbourg
  - Centre Hospitalier Du Mans, Le Mans
  - CHU de Nantes, Nantes
  - Chru Orleans, Orléans
  - CH de SAINT NAZAIRE, Saint-Nazaire
  - Hopital Foch, Suresnes
  - Chru Bretonneau - Tours, Tours
  - Centre Hospitalier Bretagne-Atlantique -Site de Vannes, Vannes